CLINICAL TRIAL: NCT04539626
Title: Estrogen Therapy in Non-severe COVID-19 Patients: Proposed Treatment Scheme in a Tertiary Hospital
Brief Title: Estrogen Therapy in Non-severe COVID-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CMN "20 de Noviembre" (Other)
Responsible Party: Principal Investigator, Alfredo Cortés Algara, Gynecology Service Member, MD, MSc, CMN "20 de Noviembre"
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03
Record Dates: First submitted 2020-09-03; First posted 2020-09-07 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Covid-19
Keywords: COVID-19; Estrogens; Severe Acute Respiratory Syndrome Coronavirus-2
MeSH Terms: conditions — COVID-19 | interventions — Estrogen Replacement Therapy; Ethinyl Estradiol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The Outcome Assessor will be an external member of the Gynecology Service, which will be blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Estrogen Therapy (Experimental): Drug: Norelgesetromin 6mg / Ethinyl estradiol 0.60mg
  Dosage form: EVRA skin patches with norelgesetromin 6mg / ethinyl estradiol 0.60mg, (1 patch will be placed every week during 21 days)
  Interventions: Drug: Estrogen Therapy
- Control Group (No Intervention): Patients who will receive conventional COVID-19 treatment

INTERVENTIONS:
Drug: Estrogen Therapy — EVRA skin patches with norelgesetromin 6mg / ethinyl estradiol 0.60mg, (1 patch will be placed every week during 21 days)
  Other Names: Norelgesetromin; Ethinyl estradiol
  Arms: Estrogen Therapy

SUMMARY:
The primary objective of this study is to evaluate the effect of additional estradiol estrogen therapy on clinical response and mortality in non-severe COVID-19 patients

DETAILED DESCRIPTION:
Actually, there is not treatment or vaccine that can prevent or control the evolution of COVID-19. The epidemiological data reported in China by the Center for Disease Control (CDC) on February 2020, reported that 87% of the patients have been adults in an age range of 30-69 years. In addition, different studies have shown that male gender are more vulnerable for the contagion of the virus (60%-80%), as well as the clinical evolution of COVID-19 (including mortality) compared to the female sex (20-40%), independently of individual such as diabetes, cardiovascular diseases, obesity, mainly.

The mechanism of SARS-CoV-2 infection has been shown to occur with the interaction of angiotensin converting enzyme 2 (ACE2), this enzyme is expressed in lungs, brain, heart, kidneys and gastrointestinal tract. Also, has been shown that older people have higher levels of ACE2 expression. Among the different molecular functions of ACE2 are the regulation of cell proliferation, cytokine production, and inflammatory response.

It has been proposed that exogenous human recombinant ACE2 could be an alternative treatment for COVID-19, however, this treatment is not yet highly available and could entail high costs. Other molecules as estrogens have been proposed in different research groups, for its capacity to increase the gene expression of ACE2/Ang 1-7. This mechanism could reduce lung and endothelial damage and coagulopathy in COVID-19 patients.

So, it is relevant to evaluate the effect of additional estradiol estrogen (as adjuvant therapeutic element) therapy on clinical response and mortality in non-severe COVID-19 patients.

A controlled clinical trial will be conducted in a tertiary hospital in Mexico City, Mexico. Participants will be divide in two groups; 1) intervention: who will receive EVRA skin patches (1 patch every week during 21 days) with norelgesetromin 6mg / ethinyl estradiol 0.60mg and 2) control: who will receive conventional treatment

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 18 years of age and female ≥ 55 years of age
* Diagnosis of positive SARS-CoV-2 infection confirmed by clinical diagnosis and / or RT-PCR test
* Hospitalized patients in acute disease* stages of the disease
* Agree to participate in the study prior to signing an informed consent.
* Patients with conventional treatment with anticoagulants (Noxaparin)

  * Acute disease: patients who are hospitalized, conscious, not intubated, with biochemical values of D-Dimer> 2, Ferritin> 1000 u.

Exclusion Criteria:

* Patients with abnormal genital bleeding
* Patients with protein C or protein S deficiency
* Patients with liver failure (cirrhosis, hepatitis C)
* Patients with history of allergic reaction to estrogens use
* Patients receiving lamotrigine therapy
* Patients with a history of breast cancer and / or endometrial cancer
* Patients with severe hypoxia at risk of acute intubation in ED
* Patients with a history of cerebrovascular history
* Male patients with testosterone treatment
* Patients with a history of myocardial infarction, who have cardiac stents and / or unstable angina pectoris
* Patients with previous hormonal treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical improve to estrogen therapy in non-severe COVID-19 patients Clinical improve to estrogen therapy in non-severe COVID-19 patients | Day 7
  * Success rate in reducing hospitalization days
  * Success rate in no oxygen therapy use (low or high-flow oxygen)
  * Success rate in no intubation and/or mechanical ventilation
  * Success rate in non mortality occurrence
Clinical improve to estrogen therapy in non-severe COVID-19 patients | Day 14
  * Success rate in reducing hospitalization days
  * Success rate in no oxygen therapy use (low or high-flow oxygen)
  * Success rate in no intubation and/or mechanical ventilation
  * Success rate in non mortality occurrence
Clinical improve to estrogen therapy in non-severe COVID-19 patients | Day 21
  * Success rate in reducing hospitalization days
  * Success rate in no oxygen therapy use (low or high-flow oxygen)
  * Success rate in no intubation and/or mechanical ventilation
  * Success rate in non mortality occurrence

SECONDARY OUTCOMES:
Symptomatic improve to estrogen therapy in non-severe COVID-19 patients | Day 7
  According to the National Committee for Epidemiological Surveillance (CONAVE) in Mexico, COVID-19 symptomatic onset rate defined as the presence of cough, fever or headache during the last 7 days, accompanied at least one of the following symptoms: dyspnea, arthralgia, myalgia, odynophagia / pharyngeal burning, rhinorrhea, conjunctivitis or chest pain.
Symptomatic improve to estrogen therapy in non-severe COVID-19 patients | Day 14
  According to the National Committee for Epidemiological Surveillance (CONAVE) in Mexico, COVID-19 symptomatic onset rate defined as the presence of cough, fever or headache during the last 7 days, accompanied at least one of the following symptoms: dyspnea, arthralgia, myalgia, odynophagia / pharyngeal burning, rhinorrhea, conjunctivitis or chest pain.
Symptomatic improve to estrogen therapy in non-severe COVID-19 patients | Day 21
  According to the National Committee for Epidemiological Surveillance (CONAVE) in Mexico, COVID-19 symptomatic onset rate defined as the presence of cough, fever or headache during the last 7 days, accompanied at least one of the following symptoms: dyspnea, arthralgia, myalgia, odynophagia / pharyngeal burning, rhinorrhea, conjunctivitis or chest pain.
Biochemical improve to estrogen therapy in non-severe COVID-19 patients | Day 7
  Percentage change from hemoglobin, hematocrit, leukocytes, erythrocytes, platelets, prothrombin, partial thromboplastin activation time, anti-thrombin activity, fibrinogen, fibrin degradation products, D-Dimer, ALT, AST, ALP, GGT, LD, albumin, cholesterol, triglycerides, HDL, LDL, C-reactive protein, estrogens and progesterone levels, pro inflammatory cytokine and nitric oxide profile.
Biochemical improve to estrogen therapy in non-severe COVID-19 patients | Day 14
  Percentage change from hemoglobin, hematocrit, leukocytes, erythrocytes, platelets, prothrombin, partial thromboplastin activation time, anti-thrombin activity, fibrinogen, fibrin degradation products, D-Dimer, ALT, AST, ALP, GGT, LD, albumin, cholesterol, triglycerides, HDL, LDL, C-reactive protein, estrogens and progesterone levels, pro inflammatory cytokine and nitric oxide profile.
Angiotensin 1-7 change after estrogen therapy in non-severe COVID-19 patientsCOVID-19 patients | Day 21
  Percentage change from Angiotensin 1-7, measured with the Human Angiotensin 1-7 ELISA kit (colorimetric) [pg/mL]

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ruz Barros, MD, Study Chair — CMN "20 de Noviembre"; Daniel Santillán Cortés, MSc, Study Chair — CMN "20 de Noviembre"; Mónica Escamilla Tilch, PhD, Study Chair — CMN "20 de Noviembre"; Juan A Pineda Juárez, PhD, Study Chair — CMN "20 de Noviembre"; Sandra Muñoz López, MD, Study Chair — CMN "20 de Noviembre"; Maricela Escarela Serrano, MD, Study Chair — CMN "20 de Noviembre"; Paul Mondragón Terán, PhD, Study Chair — CMN "20 de Noviembre"; Alberto H De la Vega Bravo, MD, Study Chair — CMN "20 de Noviembre"; Alfredo L Cortés Algara, MD, MSc, Principal Investigator — CMN "20 de Noviembre"; Samuel Reyes-Long, MSc, Study Chair — Neurociencias básicas, Instituto Nacional de Rehabilitación LGII; Cindy Bandala, MD MSc PhD, Study Chair — Neurociencias básicas, Instituto Nacional de Rehabilitación LGII; Escuela Superior de Medicina, Instituto Politécnico Nacional
Locations (1):
- CMN "20 de Noviembre", Mexico City, Benito Juárez, Mexico

IPD SHARING:
Plan to Share IPD: No